CLINICAL TRIAL: NCT06511700
Title: Implementation of the Intravitreal Injection Service Administered by Nurses: Safety and Satisfaction of the Patients Served
Brief Title: Implementation of the Intravitreal Injection Administered by Nurses
Status: Enrolling by invitation | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Susana Santos-Ruiz, Nurse, Phd Health of Science, Corporacion Parc Tauli
Other Study IDs: Intravitrial-injection2024
Record Dates: First submitted 2024-07-03; First posted 2024-07-22 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Macular Edema; Macular Degeneration; Diabetic Macular Edema
Keywords: Anti-VEGF; Intravitreal injection; Nurse; Age-related macular degeneration; Retinal vein occlusion; Diabetic macular edema; safety
MeSH Terms: conditions — Macular Edema; Macular Degeneration; Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: It is a implementation a program incorporating nurses trained in administering intravitreal injections within the functional unit of Ophthalmology following the usual technique — Internationally, some experiences demonstrate that the administration of intravitreal injections, especially by nurses trained in aseptic techniques, is feasible without compromising patient safety. Although there is already some experience in Spain, it is a new procedure within the nursing field of the Ophthalmology service for which no results have been reported.

SUMMARY:
Introduction:

Intravitreal injections involve medication administration into the eye to treat ocular diseases and protect vision. Through an injection, the medication is introduced into the vitreous cavity, an area located at the back of the eye, behind the lens. The intravitreal injection (IVI) is a minimally invasive process administered at personalized regular intervals. It is a common procedure in ophthalmology for patients who require it. International experiences demonstrate that administering intravitreal injections, especially by nurses trained in aseptic techniques, is feasible without compromising patient safety. The project presented is based on a new care model rooted in interdisciplinary collaboration in the IVI process, operationalizing it as a functional unit. This is a great opportunity to expand the scope of practice for nurses and to demonstrate, as has been done in other countries, that the same procedure currently performed by ophthalmologists can be carried out with equal safety.

Objective:

To evaluate the safety of implementing a program incorporating nurses trained in administering intravitreal injections within the functional unit of Ophthalmology at Corporation Parc Tauli.

Method:

Observational evaluation study of a care process within the functional Ophthalmology Unit, consisting of protocol application for intravitreal injection by trained nurses. Data will be collected from users receiving care from the intravitreal injection service administered by nurses under a consensual procedure within the unit. Users meeting the inclusion criteria will be eligible. Nurses will be trained internally at CCSPT by the ophthalmology team. User participation will be voluntary. Informed consent will be obtained. Data collection during the process of care will include recording selected variables. Data collection will be carried out between 2024 and 2025. The study will be conducted over 3 years.

Application and Impact:

The development of this project will allow for a safe, more efficient redistribution of our resources. The functional unit is based on a group of professionals who work and make decisions jointly. The new distribution will enable ophthalmologists to expand their availability for more complex procedures. In the future, it is expected to increase the number of users who can benefit from the IVI service and to initiate advanced competencies in the role of the ophthalmology nurse.

ELIGIBILITY:
Inclusion criteria

- People over 18 years of age who require intravitreal therapy in the ophthalmology service

Exclusion criteria

* Non-collaborators in the technique for physical, psychological or nystagmus reasons.
* Have recent evidence of blepharitis or conjunctivitis ≤15 days (ex, red eye or thick discharge) to avoid the risk of introducing infection into the eyeball.
* Suffer ischemic heart disease or recent stroke ≤3 months to avoid the risk of precipitating another vascular ischemic attack.
* With intravitreal steroid implant.
* Pregnant women: Due to the potential teratogenic effect of anti-FCEV

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People who require intravitreal therapy in the ophthalmology service of the Corporation Parc Tauli
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Complications presented during the IIV technique | In each injection during and after the procedure until the end of treatment
  Complications presented during IIV
  1.1 Pain from the placement of the blepharostat: It will be recorded as: 0=No ; 1=Yes 1.2 Pain during the injection: It will be recorded as: 0=No ; 1=Yes 1.3 Subconjunctival haemorrhage. It will be recorded as: 0=No ; 1=Yes 1.4 Post-injection ocular hypertension: It will be recorded as: 0=No ; 1=Yes 1.5 Other Complications (specified with free text)
Late post-procedure complications | In each injection during and after the procedure until the end of treatment
  Complications that arise when users leave the service. In this case, users will be asked in subsequent visits about the complications presented. They can also be reviewed from the patient's medical history.
  2.1. Pain: If pain appeared in the first 48h. It will be recorded using a Likert scale from 0 to 10, where 0 is no pain and 10 maximum pain.
  2.2 Subconjunctival haemorrhage: It will be recorded as: 0=No ; 1=Yes 2.3. Ocular hypertension: It will be recorded as: 0=No ; 1=Yes 2.4. Visual ability to perform AVDs: To assess the current state of their vision, we will be asked if they currently notice that they can do their usual activities better or not. It will be recorded as: 0= Worsening ; 1= Maintenance; 2= Improvement 2.5. Visit to the emergency room (or ophthalmology service) for problems after the IIV. It will be recorded as: 0=No ; 1=Yes, and free text that answer to what problem did they present.

SECONDARY OUTCOMES:
Sociodemographic variables | At the beginning of treatment
  Years old, gender, family coexistence
Date of treatment indication | At the beginning of treatment
  This is the date the procedure was indicated. It will be recorded as YYYY/MM/DD
Ocular Diagnosis | At the beginning of treatment
  The main diagnosis that makes IIV indicated. It will be recorded as free text.
Ocular comorbidity | At the beginning of treatment
  Presence of another associated eye pathologies. It will be recorded as free text.
Previous experience | At the beginning of treatment
  We will ask if the patient had received IIV therapy from an ophthalmologist some time ago. If so, it don't need to ask again.
  It will be recorded as: 0= No; 1=Yes
Companion | In each injection until the end of the treatment
  Family presence at the session. It will be recorded as: 0= alone; 1=Accompanied
Visit to the ophthalmologist between therapies | In each injection until the end of the treatment
  Inquiry about the patient's visit ophthalmologist between IIV sessions. Cycles of a specific number of sessions are usually scheduled and then they are visited at the ophthalmology consultation to review the effectiveness and maintenance of the treatment, being able to change the type of drug.
  It will be recorded as: 0=No; 1=Yes
Anxiety level | In each injection until the end of the treatment
  Anxiety presented before the procedure. It will be evaluated using a Likert scale from 0 to 10, where 0 is minimum anxiety and 10 maximum anxiety.
Treated eye | In each injection until the end of the treatment
  Registration of the eye that receiving the IIV: 0=right, 1=left, 2=both.
Ophthalmologist visit during the session | In each injection until the end of the treatment
  The responsible ophthalmologist must be available during IIV session for any questions that may arise.
  If any query has to be made it will be recorded: 0=No; =Yes. If so, the reason must be specified (free text).
IVI Medication | In each injection until the end of the treatment
  Record of intravitreal medication administered. Record: 1 = Aflibercept (EYLEA®) ; 2= Bevacizumab (AVASTIN®); 3= Ranibizumab (LUCENTIS®); 4=Intravitreal Dexamethasone (OZURDEX®) 5= Others (specify). Drugs 1, 2 and 3 are drugs that inhibit vascular endothelial growth factor (anti-VEGF) and will be the two that will initially begin IIV for the nurses. On the 4th, for the present presentation and special administrative provision, initially excluded from being administered by nursing, it will be administered in three sessions by ophthalmologists.
  During 2024, the addition of a new Anti-FEVG to the CCSPT, Faricimab (VABYSMO®), is planned, which is expected to be important from a quantitative point of view in the total IIV.
Patient Pain | In each injection until the end of the treatment
  Pain that is present during IIV. It will be recorded using a Likert scale from 0 to 10, 0 no pain and 10 the most pain.
Patient Satisfaction | In each injection until the end of the treatment
  No validated questionnaire has been found in the literature to assess patient satisfaction with intravitreal therapy. Therefore, the criteria used by the study by Austen et al will be used in the consultation.
  They developed a simple satisfaction questionnaire in accordance with the guidelines for measuring the quality of health services. It consists of 2 questions with a Likert scale from 1 to 5, one related to satisfaction and the other to trust.
  In the case of answering with a low score, they are accompanied by a clarification question to improve these aspects (free text).

CONTACTS AND LOCATIONS:
Locations (1):
- Corporation Parc Tauli, Sabadell, Barcelona, Spain